CLINICAL TRIAL: NCT05004285
Title: A Multi Center, Non-randomized, Open, Phase 3 Study to Evaluate the Clinical Usefulness of [F-18]Florastamin PET/CT Imaging Diagnosis Compared to MRI Diagnosis in Prostate Cancer Risk Groups
Brief Title: Evaluate the Clinical Usefulness of [F-18]Florastamin PET/CT Imaging Diagnosis Compared to MRI Diagnosis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: FutureChem (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Protocol FC303-3
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: High Risk Prostate Carcinoma
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: compare PET/CT Imaging Diagnosis with MRI Diagnosis for one subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI / [F-18]Florastamin (Other): MRI and [F-18]Florastamin PET/CT are performed for each subject.
  Interventions: Drug: [F-18]Florastamin

INTERVENTIONS:
Drug: [F-18]Florastamin — A single dose of [F-18]Florastamin at 10 ± 1 mCi is IV administered at Visit 2, and [F-18]Florastamin PET/CT images are obtained from the head to thigh after 110 ± 10 minutes.

SUMMARY:
Only in subjects who satisfy the inclusion/exclusion criteria, a single dose of [F-18]Florastamin at 10 ± 1 mCi is IV administered at Visit 2, and [F-18]Florastamin PET/CT images are obtained from the head to thigh after 110 ± 10 minutes.

DETAILED DESCRIPTION:
Once a subject provides voluntary written consent on participation in this study, the investigator conducts screening of the subject. Subsequently, MRI and [F-18]Florastamin PET/CT are performed for each patient, only for those who satisfy the inclusion/exclusion criteria. For MRI at Visit 2, routine MRI, as implemented in the Urology Department, is performed in the abdomen and pelvis. On the date of or within 7 days after MRI, a single dose of [F-18]Florastamin at 10 ± 1 mCi is IV administered to a subject, and PET/CT images are obtained from the head to thigh after 110 ± 10 minutes (care should be taken to prevent extravasation of the radiopharmaceutical product). At Visit 3, the principal investigator or a treating doctor as delegated by the principal investigator conducts the template prostate-mapping (TPM) biopsy in at least the Modified Barzell 20-zone using the standard template. After general anesthesia or spinal anesthesia, the tissue is collected by horizontally sticking a histological needle through the perineum, and the process can be performed as in-patient, at the discretion of the investigator.

The MRI finding is determined positive for a lesion with the PI-RADS score of 3 or higher, and the [F-18]Florastamin PET/CT finding is considered positive for the focal uptake higher than the background level and unrelated with the physiologic uptake or known pitfall.

MRI and [F-18]Florastamin PET/CT images are sent to the central reading institution, Seoul St. Mary's Hospital, after blinding for the study information. Suspected sites on MRI are evaluated at the Seoul St. Mary's Hospital Radiology Department, and the suspected sites on [F-18]Florastamin PET/CT are assessed at the Seoul St. Mary's Hospital Nuclear Medicine Department. Note that the [F-18]Florastamin PET/CT rater would participate in the assessment after undergoing sufficient training with [F-18]Florastamin PET/CT images from a Phase 1 study of the same product.

A pathologist at each center will conduct diagnosis of prostate cancer for TPM biopsy samples from the entire prostate volume. Target biopsy of MRI and [F-18]Florastamin PET/CT will not be performed. By comparing confirmed sites from each imaging diagnosis method and positive/negative results for prostate cancer from TPM biopsy diagnosis, the proportions of True Positive (TP), False Positive (FP), True Negative (TN), False Negative (FN) will be analyzed and the sensitivity, specificity, negative predictive value, positive predictive value, and diagnostic accuracy will be compared using a 2x2 contingency table.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men aged at least 20 years determined to be at the high risk of prostate cancer based on screening diagnosis performed at the Urology Department (Patients who require prostate histology due to abnormal digital rectal examination (DRE) or abnormal PSA levels, etc., and have a palpable node during DRE or satisfy PSA>3.0 ng/mL)
2. Subjects who were not previously diagnosed with prostate cancer at the time of screening
3. Subjects who can conduct prostate histology
4. Subjects with the ECOG Performance score of ≤2 at screening
5. Subjects who satisfy the following conditions for hematology, kidney function test and liver function test

   ① Platelets > 50,000/mm3

   ② BUN and serum creatinine < 1.5 x upper limit of normal (ULN)

   ③ AST and ALT < 2.5 x upper limit of normal (ULN)

   ④ PT (INR) or aPTT < 1.5 x upper limit of normal (ULN)
6. Subjects who were fully informed by the investigator about the objectives, details of the study and characteristics of the study drug, etc. during the screening visit and provide voluntary written consent to take part in this study

Exclusion Criteria:

1. Subjects who were previously diagnosed with prostate cancer
2. Subjects with a history of acute urinary retention, urinary tract infection or other urinary infection within 4 weeks of screening
3. Subjects who conducted cystoscopy, urethral catheter procedure or colonoscopy within 4 weeks of screening
4. Subjects who conducted prostate histology or prostate surgery (other than treatment for prostate hyperplasia or bladder outlet obstruction) or androgen deprivation therapy (ADT) within 1 year of screening
5. Subjects who received 5-alpha reductase inhibitors within 3 months of screening or currently on them at screening
6. Subjects with hypersensitivity to any component of the radiopharmaceutical product
7. Subjects determined by the investigator to have difficulty in conducting the study due to serious medical disease
8. Subjects determined by the investigator to have difficulty in lying still for 30-60 minutes in a supine position for radiography (CT, MRI, etc.) (example: panic disorder) or have psychiatric disorder causing difficulty in imaging
9. Subjects who are planned to administer contraindicated concomitant medication (antiplatelet agents/anticoagulants, thrombolytics or circulatory improvement agents) between 5 days before biopsy and [Visit 3 + 3D]
10. Subjects who are otherwise determined to be ineligible to take part in this study at the medical discretion of the investigator

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients aged 20 years or older.
Enrollment: 398 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity and specificity analyzed for patients based on histological findings | MRI and PET/CT conduct at V2(0 day), TPM Biopsy conduct at V3(V2+1~14 day).
  For the sensitivity and specificity analyzed for patients of MRI diagnostic imaging and PET/CT diagnostic imaging based on histological findings, present the frequency, percentage and corresponding 95% confidence interval for each group, and conduct the McNemar's test for between-group difference. If the p-value from the McNemar's test is <0.05 for both sensitivity and specificity, superiority of PET/CT diagnostic imaging to MRI diagnostic imaging is declared.

SECONDARY OUTCOMES:
Diagnostic sensitivity analyzed for lesions based on histological findings | MRI and PET/CT conduct at V2(0 day), TPM Biopsy conduct at V3(V2+1~14 day).
  For the following endpoints, present the frequency, percentage and corresponding 95% confidence interval for each group, and conduct the McNemar's test for between-group difference
Diagnostic specificity analyzed for lesions based on histological findings | MRI and PET/CT conduct at V2(0 day), TPM Biopsy conduct at V3(V2+1~14 day).
  For the following endpoints, present the frequency, percentage and corresponding 95% confidence interval for each group, and conduct the McNemar's test for between-group difference
Negative predictive value of diagnosis analyzed for patients based on histological findings | MRI and PET/CT conduct at V2(0 day), TPM Biopsy conduct at V3(V2+1~14 day).
  For the following endpoints, present the frequency, percentage and corresponding 95% confidence interval for each group, and test for the between-group difference with generalized score statistics
Positive predictive value of diagnosis analyzed for patients based on histological findings | MRI and PET/CT conduct at V2(0 day), TPM Biopsy conduct at V3(V2+1~14 day).
  For the following endpoints, present the frequency, percentage and corresponding 95% confidence interval for each group, and test for the between-group difference with generalized score statistics.
Negative predictive value of diagnosis analyzed for lesions based on histological findings | MRI and PET/CT conduct at V2(0 day), TPM Biopsy conduct at V3(V2+1~14 day).
  For the following endpoints, present the frequency, percentage and corresponding 95% confidence interval for each group, and test for the between-group difference with generalized score statistics.
Positive predictive value of diagnosis analyzed for lesions based on histological findings | MRI and PET/CT conduct at V2(0 day), TPM Biopsy conduct at V3(V2+1~14 day).
  For the following endpoints, present the frequency, percentage and corresponding 95% confidence interval for each group, and test for the between-group difference with generalized score statistics.
Diagnostic accuracy analyzed for patients based on histological findings | MRI and PET/CT conduct at V2(0 day), TPM Biopsy conduct at V3(V2+1~14 day).
  For the following endpoints, present the frequency, percentage and corresponding 95% confidence interval for each group, and conduct the McNemar's test for between-group difference
Diagnostic accuracy analyzed for lesions based on histological findings | MRI and PET/CT conduct at V2(0 day), TPM Biopsy conduct at V3(V2+1~14 day).
  For the following endpoints, present the frequency, percentage and corresponding 95% confidence interval for each group, and conduct the McNemar's test for between-group difference
Proportion of subjects who can be excluded from histology among those who are determined to be positive from MRI (PI-RADS ≥3) diagnosis but negative from [F-18]Florastamin PET/CT diagnosis based on histological findings | MRI and PET/CT conduct at V2(0 day), TPM Biopsy conduct at V3(V2+1~14 day).
  Present the proportion and corresponding 95% confidence interval of subjects who can be excluded from histology among those who are determined to be positive from MRI (PI-RADS ≥3) diagnosis but negative from [F-18]Florastamin PET/CT diagnosis based on histological findings

CONTACTS AND LOCATIONS:
Overall Officials: Ji Youl Lee, Ph.D, Principal Investigator — The Catholic University of Korea
Locations (5):
- South Korea (5):
  - National Cancer Center, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catalona WJ, Partin AW, Slawin KM, Brawer MK, Flanigan RC, Patel A, Richie JP, deKernion JB, Walsh PC, Scardino PT, Lange PH, Subong EN, Parson RE, Gasior GH, Loveland KG, Southwick PC. Use of the percentage of free prostate-specific antigen to enhance differentiation of prostate cancer from benign prostatic disease: a prospective multicenter clinical trial. JAMA. 1998 May 20;279(19):1542-7. doi: 10.1001/jama.279.19.1542. PMID 9605898
- [Background] Park HK, Hong SK, Byun SS, Lee SE. T1c prostate cancer detection rate and pathologic characteristics: comparison between patients with serum prostate-specific antigen range of 3.0 to 4.0 ng/mL and 4.1 to 10.0 ng/mL in Korean population. Urology. 2006 Jul;68(1):85-8. doi: 10.1016/j.urology.2006.01.067. Epub 2006 Jun 27. PMID 16806412
- [Background] Johnson DC, Raman SS, Mirak SA, Kwan L, Bajgiran AM, Hsu W, Maehara CK, Ahuja P, Faiena I, Pooli A, Salmasi A, Sisk A, Felker ER, Lu DSK, Reiter RE. Detection of Individual Prostate Cancer Foci via Multiparametric Magnetic Resonance Imaging. Eur Urol. 2019 May;75(5):712-720. doi: 10.1016/j.eururo.2018.11.031. Epub 2018 Dec 1. PMID 30509763
- [Background] Hofman MS, Murphy DG, Williams SG, Nzenza T, Herschtal A, Lourenco RA, Bailey DL, Budd R, Hicks RJ, Francis RJ, Lawrentschuk N. A prospective randomized multicentre study of the impact of gallium-68 prostate-specific membrane antigen (PSMA) PET/CT imaging for staging high-risk prostate cancer prior to curative-intent surgery or radiotherapy (proPSMA study): clinical trial protocol. BJU Int. 2018 Nov;122(5):783-793. doi: 10.1111/bju.14374. Epub 2018 Jun 3. PMID 29726071
- [Background] Chang SS. Overview of prostate-specific membrane antigen. Rev Urol. 2004;6 Suppl 10(Suppl 10):S13-8. PMID 16985927
- [Background] Szabo Z, Mena E, Rowe SP, Plyku D, Nidal R, Eisenberger MA, Antonarakis ES, Fan H, Dannals RF, Chen Y, Mease RC, Vranesic M, Bhatnagar A, Sgouros G, Cho SY, Pomper MG. Initial Evaluation of [(18)F]DCFPyL for Prostate-Specific Membrane Antigen (PSMA)-Targeted PET Imaging of Prostate Cancer. Mol Imaging Biol. 2015 Aug;17(4):565-74. doi: 10.1007/s11307-015-0850-8. PMID 25896814
- [Background] Maurer T, Eiber M, Schwaiger M, Gschwend JE. Current use of PSMA-PET in prostate cancer management. Nat Rev Urol. 2016 Apr;13(4):226-35. doi: 10.1038/nrurol.2016.26. Epub 2016 Feb 23. PMID 26902337
- [Background] Rhee H, Thomas P, Shepherd B, Gustafson S, Vela I, Russell PJ, Nelson C, Chung E, Wood G, Malone G, Wood S, Heathcote P. Prostate Specific Membrane Antigen Positron Emission Tomography May Improve the Diagnostic Accuracy of Multiparametric Magnetic Resonance Imaging in Localized Prostate Cancer. J Urol. 2016 Oct;196(4):1261-7. doi: 10.1016/j.juro.2016.02.3000. Epub 2016 May 21. PMID 27220897
- [Background] Lee I, Lim I, Byun BH, Kim BI, Choi CW, Woo SK, Lee KC, Kang JH, Kil HS, Park C, Chi DY, Park J, Song K, Lim SM. A microdose clinical trial to evaluate [18F]Florastamin as a positron emission tomography imaging agent in patients with prostate cancer. Eur J Nucl Med Mol Imaging. 2021 Jan;48(1):95-102. doi: 10.1007/s00259-020-04883-y. Epub 2020 May 26. PMID 32458006
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Valerio M, Anele C, Charman SC, van der Meulen J, Freeman A, Jameson C, Singh PB, Emberton M, Ahmed HU. Transperineal template prostate-mapping biopsies: an evaluation of different protocols in the detection of clinically significant prostate cancer. BJU Int. 2016 Sep;118(3):384-90. doi: 10.1111/bju.13306. Epub 2015 Sep 25. PMID 26332050
- [Background] Weinreb JC, Barentsz JO, Choyke PL, Cornud F, Haider MA, Macura KJ, Margolis D, Schnall MD, Shtern F, Tempany CM, Thoeny HC, Verma S. PI-RADS Prostate Imaging - Reporting and Data System: 2015, Version 2. Eur Urol. 2016 Jan;69(1):16-40. doi: 10.1016/j.eururo.2015.08.052. Epub 2015 Oct 1. PMID 26427566
- [Background] Leisenring W, Alonzo T, Pepe MS. Comparisons of predictive values of binary medical diagnostic tests for paired designs. Biometrics. 2000 Jun;56(2):345-51. doi: 10.1111/j.0006-341x.2000.00345.x. PMID 10877288
- [Background] Wang W, Davis CS, Soong SJ. Comparison of predictive values of two diagnostic tests from the same sample of subjects using weighted least squares. Stat Med. 2006 Jul 15;25(13):2215-29. doi: 10.1002/sim.2332. PMID 16220470
- [Background] Li J, Fine J. On sample size for sensitivity and specificity in prospective diagnostic accuracy studies. Stat Med. 2004 Aug 30;23(16):2537-50. doi: 10.1002/sim.1836. PMID 15287083
- [Background] Jia Y, Zhu LY, Xian YX, Sun XQ, Gao JG, Zhang XH, Hou SC, Zhang CC, Liu ZX. Detection rate of prostate cancer following biopsy among the northern Han Chinese population: a single-center retrospective study of 1022 cases. World J Surg Oncol. 2017 Aug 29;15(1):165. doi: 10.1186/s12957-017-1238-9. PMID 28851376
- See also: Prostate Specific Antigen (PSA) Test, Results, Levels & Ranges — https://www.medicinenet.com/prostate_specific_antigen/article.htm